CLINICAL TRIAL: NCT06450678
Title: Use of a Physiotherapy Assessment to Predict Extubation Failure in Mechanically Ventilated Patients: the EPIC Assessment
Acronym: PREDEXTUB
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231743; 2023-A01734-41 (Other: ID-RCB)
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Mechanical Ventilator Weaning; Mechanical Ventilation
Keywords: ICU; extubation failure; predictive factors; physiotherapist

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with mechanical ventilation: Adult patients admitted to intensive care with mechanical ventilation for more than 48 hours

SUMMARY:
"Weaning from mechanical ventilation is a crucial step in the intensive care unit. Several factors complicate weaning and increase the risk of failure. To predict the success of extubation, the spontaneous ventilation test (T-Tube) remains essential. Despite this, the failure rate is around 10-20%.

Failed extubation is not without consequences, since it increases the risk of pneumopathy and mortality. It therefore seems essential to identify potential extubation failures using effective predictive criteria. Several of these predictive criteria have been studied separately in the literature, but are still not widely used in practice. Many studies have sought to identify these predictive criteria, without actually linking them. However, when combined in a single assessment prior to extubation, they could represent a reliable prediction and decision-making aid.

In the intensive care unit at Hôpital Bichat Claude Bernard, a team of physiotherapists dedicated solely to this unit carries out a routine EPIC Assessment, combining several criteria, some of which have individually demonstrated their reliability in predicting extubation outcome. Physiotherapists are health professionals working as part of the intensive care team, and are well versed in issues relating to bronchial congestion, respiratory function and muscle strength, whether for breathing or locomotion. Similarly, their involvement in issues relating to swallowing disorders acquired in intensive care gives them an overall view of the patient's ability to protect his or her airway post-extubation. The EPIC Assessment has been designed by them to address these issues. With the help of this assessment, and by following the cut-offs of the various criteria, they link the different criteria making up the EPIC Assessment and communicate a ""favorable"" or ""unfavorable"" opinion for extubation.

Our hypothesis is that the EPIC Assessment is, in addition to its interpretation by physiotherapists, a reliable tool for predicting the outcome of extubation."

DETAILED DESCRIPTION:
Adult patients admitted to the ICU and placed on invasive mechanical ventilation for more than 48 hours will be screened by the investigators (physiotherapists in conjunction with a doctor).

The spontaneous ventilation test will be carried out in the T-Tube, on the basis of a medical decision and within the framework of care, if the patients meet the weaning conditions:

* No sedation
* No inotropes or vasopressors
* Consistent response to simple commands
* FiO2 < 50%
* PEEP < 5 cmH2O

The criteria for a successful T-Tube test are:

* FR < 35 cycles/min
* SpO2 > 90%,
* Variation of less than 20% in FR or systolic blood pressure,
* No sweating, agitation or vigilance disorders.

Inclusion of patients by investigators after a successful spontaneous ventilation test.

Data will be collected describing the characteristics of patients on the day of their T-Tube test, and will also list the various risk factors for extubation failure already known in the literature, in order to avoid confounding bias

EPIC Assessment by physiotherapists: Within 30 minutes of a successful spontaneous ventilation test, the physiotherapists are called in by the nursing team to carry out the EPIC Assessment. This assessment takes the form of a table containing the following criteria:

* Glasgow Coma Scale (GCS): X < 11 ≤ O
* Rapid Shallow Breathing Index (RSBI): X ≤ 75 < O
* Maximum Inspiratory Pressure (MIP): X < l-25l < O
* Peak Expiratory Flow (PEF): X < l-60l < O
* Bronchial congestion: X = "++" and "+++"; O = "+" and "Ø"
* Salivary stasis: X = "++" and "+++"; O = "+" and "Ø".
* Orofacial motricity: X = Incomplete and O = Complete
* Cervical spine flexion: X = Impossible and O = Possible
* Nausea reflex: X = Absent and O = Present on at least one side.
* Medical Research Council (MRC): X < 36 and O > 36.

The patient is placed in a semi-sitting position, having been lifted into bed beforehand.

The physiotherapist first takes information about the starting conditions, then decreases the Inspiratory Pressure (IP) to 7 and the Positive Expiratory Pressure (PEP) to 0.

Each criterion is then assessed by the physiotherapist with the patient's participation. The cut-offs described in the literature are taken into account to validate each criterion: an "X" sign predicts extubation failure, an "O" sign predicts extubation success.

Inter-rater reproducibility study: the EPIC grids will be reviewed at the end of the research by a physiotherapist who has not carried out this EPIC, who will be responsible for giving a "favorable" or "unfavorable" opinion based on the results of the EPIC assessment (opinion not taken into account for the extubation decision - for reproducibility analysis only).

Binary global assessment: "favorable" or "unfavorable" opinion, issued collectively by the entire team in charge of the patient (physiotherapist, senior doctor, junior doctor (intern), state-registered nurse, nursing auxiliary).

Extubation decision: taken by the doctor after the spontaneous ventilation test and communication by the physiotherapists of their favorable or unfavorable opinion. Participation in the research will not affect patient management. A patient who has not been extubated will be reassessed according to the care plan in the following days (new spontaneous ventilation test, new EPIC assessment).

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Admitted to intensive care and placed on invasive mechanical ventilation for more than 48 hours
* Having passed a T-Tube spontaneous ventilation test < 24h

Exclusion Criteria:

* Tracheostomized patient
* Severe psychiatric pathology or cognitive disorders
* Uncooperative patient
* Patient under therapeutic restriction (terminal extubation)
* Patient who has already participated in research
* Patient or close relative (if patient not able) opposed to research
* No relative if patient unable to receive information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to intensive care and placed on invasive mechanical ventilation for more than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
extubation failure rate | day 7 after extubation

SECONDARY OUTCOMES:
extubation failure rate | 48h after extubation
extubation failure rate | 72h after extubation
Length of stay in post-extubation intensive care unit | 1 month
Total length of hospital stay post-extubation | 1 month
in-hospital death rate | 1 month
Binary global assessment: "favorable" or "unfavorable" opinion on extubation, given collectively by the caregivers in charge of the patient (physiotherapist, senior physician, junior physician (intern), state-registered nurse, nursing auxiliary). | at extubation
"Favourable" or "unfavourable" rating by two assessors (physiotherapists) blind to the other assessor's rating | at extubation
Medical decision to extubate (or not) the patient following a positive (or negative) opinion from the physiotherapist | at extubation
Glasgow Coma Scale | The intubated patient's GCS does not take into account the verbal component, as the patient is unable to speak.
  before extubation
Rapid Shallow Breathing Index | before extubation
  "RSBI is performed within the first few minutes of the assessment by the physiotherapists.
  On the ventilator, the mean tidal volumes in one minute are taken, and the respiratory rate is also measured."
Measurement of Maximum Inspiratory Pressure | before extubation
  MIP is obtained on the ventilator, using the dedicated function. The physiotherapist applies a 7-second expiratory pause at the end of exhalation and asks the patient to inhale. This maneuver is performed 3 times, and the best of the three values is taken into account.
Measurement of Peak Expiratory Flow | before extubation
Measurement of Bronchial congestion | before extubation
  The patient's state of congestion is rated by the physiotherapist, taking into account the patient's state of congestion over the 24 hours (assessed by the nurses and orderlies during rounds and noted on the sign) and according to the aspirations performed.
Measurement of Salivary stasis | before extubation
  The patient's salivary stasis status is rated by the physiotherapist, taking into account the patient's salivary stasis over the 24 hours (assessed by the nurses and orderlies during rounds and noted on the sign) and according to the aspirations performed.
Measurement of Orofacial motor control | before extubation
  The patient is asked to: open the mouth; stick out the tongue and move it to the right and left; smile.
Measurement of Cervical spine flexion | before extubation
  The patient is asked to lift his or her head from the pillow and to hold it there.
Measurement of Nausea reflex | before extubation
  The physiotherapist inserts a 10ml syringe between the patient's teeth, and stimulates the right and left pillars of the pharynx with a finger. A contraction of the pharynx accompanied by a sensation of discomfort on the part of the patient validates the presence of the nausea reflex
Medical Research Council | before extubation
Laryngeal lift | before extubation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine SHENOUDA, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat - Claude Bernard Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided